CLINICAL TRIAL: NCT04283513
Title: Treatment Protocol for Adults With Hemorrhagic Fever With Renal Syndrome (HFRS) With Intravenous (IV) Ribavirin
Brief Title: Treatment of Hemorrhagic Fever With Ribavirin
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-16-01
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Hemorrhagic Fever
Keywords: Hemmorrhagic Fever; Ribavirin
MeSH Terms: conditions — Hemorrhagic Fevers, Viral | interventions — Ribavirin

STUDY DESIGN:
Intervention Model Description: This protocol is an open-label, single-arm, multisite protocol to provide IV ribavirin treatment to patients with probable or suspected case of Hemorrhagic Fever with Renal Syndrome (HFRS).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Efficacy of IV Ribavirin (Experimental): The proposed clinical dose is based on drug dosage used in the HFRS clinical trial in China that demonstrated efficacy: Loading dose, 33 mg/kg (maximum dose: 2.64 g), followed by a dose of 16 mg/kg (maximum dose: 1.28 g) every 6 hours for the first 4 days (15 doses), and 8 mg/kg (maximum dose: 0.64 g) every 8 hours for the subsequent 3 days (9 doses).
  Interventions: Drug: Virazole

INTERVENTIONS:
Drug: Virazole — Virazole (Ribavirin), USP Injection 0.1 g/mL in a phosphate buffer solution. Each vial contains 1.2 g of Ribavirin in 12 mL
  Other Names: IV Ribavirin

SUMMARY:
Multisite protocol to provide IV Ribavirin treatment to patients with probable or suspected case of Hemorrhagic Fever with Renal Syndrome (HFRS)

DETAILED DESCRIPTION:
This protocol is an open-label, single-arm, multisite protocol to provide IV ribavirin treatment to patients with probable or suspected case of HFRS. Individuals with a tentative diagnosis of HFRS will be admitted to the MTF and treated for up to 7 days with doses of IV ribavirin.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet all of the following criteria to be included in the study:

* Meets the protocol case definition for a probable or suspected case (see Section 8.5.2 and Section 8.5.3)
* Has read and signed the Informed Consent.
* Must be Department of Defense (DoD)-affiliated personnel including active and reserve component service members, US civilian employees, contractors, other US Personnel, and dependents as well as allied military forces and local nationals who have been granted access to the medical facility.
* Is at least 18 years of age (17, if active military) and not greater than 65 years of age.
* Agrees to have a blood sample drawn and a type and cross-match ordered for transfusion.
* Agrees to collection of required specimens.
* Agrees to report any adverse events (AEs) for the duration of the patient's treatment protocol participation.
* Agrees to follow-up visits and to donate blood and urine specimens at Day 10, Day 14, and once between Days 28 and 60 after the first dose of IV ribavirin and to all follow-up visits for anemia or other medical conditions as required by the attending physician.
* Has a hemoglobin of 10 g/dL or higher before starting IV ribavirin.
* Women who are breastfeeding agree to discontinue breastfeeding during treatment with IV ribavirin and during the 7-month post-treatment period.
* Woman of childbearing potential must have a negative pregnancy test within 24 hours before starting treatment and agrees not to become pregnant during treatment and for 7 months after receiving IV ribavirin. Treatment will be a maximum of 25 doses given over a 1 week time period. At least 2 reliable forms of effective contraception, including 1 barrier method, must be utilized during treatment and during the 7 months post treatment period.(See Section 12.1.6 Pregnancy)
* Male subjects agree not to have intercourse with pregnant women during treatment and for 7 months after receiving IV ribavirin, and take precautions to avoid producing pregnancies in female partners during and for 7 months after receiving ribavirin. Treatment will be a maximum of 25 doses given over a 1 week time period. At least 2 reliable forms of effective contraception, including 1 barrier method, must be utilized during the treatment and during the 7 month post-treatment period (See Section 12.1.6 Pregnancy). Their female partner should use a highly effective contraceptive method (see Section 12.1.6). They agree to use a male condom plus an additional method with a failure rate of < 1% per year).

Exclusion Criteria:

Individual will not be enrolled in the protocol if they meet any of the following criteria:

* Has a known intolerance to ribavirin.
* Is irreversibly ill on presentation, as defined by presence of profound shock, which does not respond to supportive therapy within 3 hours after admission.
* Has a positive pregnancy test.
* Has an estimated creatinine clearance < 20 mL/minute
* Is receiving renal dialysis.
* Has a history of hemoglobinopathies (ie, sickle-cell anemia or thalassemia major).
* Has a history of autoimmune hepatitis.
* Has a hemoglobin less than 10 g/dL that cannot be corrected to ≥ 10 g/dL before initiation of IV ribavirin.
* Has a New York Heart Association Cardiac functional capacity of Class II or greater for atherosclerotic heart diseases (ASHD) and congestive heart failure (CHF). Class II ASHD or greater includes angina that occurs at rest, with daily activities, and/or with slightly more prolonged or with slightly more vigorous activity than usual. Class II CHF or greater includes CHF resulting in mild symptoms with ordinary physical activity, or marked or severe limitations of activity [See Appendix B for New York Heart Association Functional Classification of Angina and CHF].
* Has known cardiac conduction defects that may predispose the patient to arrhythmias such as WPW; or a history of bradyarrhythmias, such as second or third degree heart block or sick sinus syndrome and no pacemaker
* Has a sinus bradycardia of less than 40 beats per minute (or sinus bradycardia less than 50 beats per minute if the individual is not known to have a low resting heart rate related to physical conditioning).
* Is currently being treated with didanosine (ddI) or azathioprine. DdI and azathioprine must be discontinued before starting IV ribavirin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Reduction in Mortality with IV Ribavirin at 10days | 10 Days (+/-1)
  Measuring the treatment effectiveness of the injected IV Ribavirin by the reduction of mortality and reported serious adverse events at the 10 days interval.
Reduction in Mortality with IV Ribavirin at 14days | 14 Days (+/-2)
  Measuring the treatment effectiveness of the injected IV Ribavirin by the reduction of mortality and reported serious adverse events at the 14 days interval.
Reduction in Mortality with IV Ribavirin at 28-60days | 28-60 Days
  Measuring the treatment effectiveness of the injected IV Ribavirin by the reduction of mortality and reported serious adverse events at the 28-60 days interval.

SECONDARY OUTCOMES:
Reported Adverse Events | 0-60 days
  Number of patient reported Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Landstuhl Regional Medical Center, Landstuhl, Germany

IPD SHARING:
Plan to Share IPD: No